CLINICAL TRIAL: NCT06512142
Title: Using Artificial Intelligence for the Detection of Respiratory Diseases Associated With Pollution
Acronym: SmartLungs
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Responsible Party: Principal Investigator, Ana Adriana Trusculescu, Dr., University of Medicine and Pharmacy "Victor Babes" Timisoara
Other Study IDs: PostdocTrusculescu/11.2023
Record Dates: First submitted 2024-07-15; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: COPD Asthma; Lung Neoplasm; Emphysema
Keywords: complex networks; lung imaging; spectral analysis; geolocation
MeSH Terms: conditions — Lung Neoplasms; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Generating a picture at the city level, through geospatial and temporal grouping a lung diseases associated or exacerbated by pollution (COPD, AB and neoplasm pulmonary or pleural) and correlating this data with pollution data.

Development of an accurate and prognostic HRCT imaging diagnostic tool, computer assisted in the mentioned pathology, by generating an algorithm capable of to detect early the follow-up tomographic imaging lesions, as well as to evaluate objective their speed of evolution.

Validation of the proposed algorithm by comparison with medical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with COPD and/or asthma and/or pulmonary neoplasm and/or secondary pulmonary, pleural or mediastinal determinations, suspected or confirmed, according to ICD-10.
* Patients will be included regardless of the type of hospitalization, continuous or day.
* The existence of freely expressed consent, carried out according to Ethics standards professional (from the observation sheet).

For stage 2

* The use of HRCT images, in DICOM format, with a maximum cup thickness of 1.5 mm and with an average of 250 cups; no image acquisition errors;
* Imaging monitoring at a time interval;.
* Respiratory function evaluation data available: spirometry +/- the factor of gaseous diffusion (DLco);

Exclusion Criteria:

For both stages:

- Patients who do not have a stable real domicile (eg social cases) or are not from the Timis county

For stage 2

* Patients who do not have HRCT images available or cannot be followed.
* Patients who have insufficient quality HRCT images.
* Patients who have a history of lung surgery.
* Patients who have a history of allergies to contrast agents used in imaging HRCT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary specialized Victor Babes Respiratory Hospital patients
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between lung diseases and pollution | December 2023 - December 2024
  Establishing the relationship between the incidence and exacerbation of lung diseases (COPD, acute bronchitis, and pulmonary or pleural neoplasms) and pollution levels through geospatial and temporal analysis at the city /county level
Development of a diagnostic algorithm | September 2024 - March 2024
  Creating an accurate, computer-assisted HRCT imaging diagnostic tool designed to detect early tomographic lesions and evaluate the progression speed of these lesions in patients with the mentioned pathologies.

CONTACTS AND LOCATIONS:
Locations (1):
- "Victor Babes" University Hospital, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No